CLINICAL TRIAL: NCT06910241
Title: Lidocaine Versus Diphenhydramine to Achieve Local Anesthesia for Laceration Repairs
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Florida Atlantic University (Other)
Collaborators: Baptist Health South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2195722
Record Dates: First submitted 2025-04-02; First posted 2025-04-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Laceration of Skin
MeSH Terms: interventions — Lidocaine; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Active Comparator)
  Interventions: Drug: Lidocaine
- Diphenhydramine (Experimental)
  Interventions: Drug: Diphenhydramine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine local infiltration
  Arms: Lidocaine
Drug: Diphenhydramine — Diphenhydramine local infiltration
  Arms: Diphenhydramine

SUMMARY:
Diphenhydramine, when injected locally, has been shown to achieve a certain level of local anesthesia. It has been documented for use in simple bedside procedures, however there is a gap in knowledge in its comparison to lidocaine. The purpose of the study is to determine if local infiltration of diphenhydramine is noninferior to the use of lidocaine 1% when trying to achieve local anesthesia for simple laceration repair. Patients who present to the emergency department with a simple laceration will be enrolled in the study. Patients will be evaluated for the pain of the injection as well as the pain of the laceration repair procedure post injection.

ELIGIBILITY:
Inclusion Criteria:

* Lacerations requiring one layer of sutures
* Lacerations appropriate for repair by emergency physicians

Exclusion Criteria:

* Active bleeding from laceration
* Complex lacerations requiring multiple layers
* Lacerations to be repaired by a specialist service
* Patients with allergies to either diphenhydramine or lidocaine
* Laceration repairs would benefit from the use of epinephrine as an additive to the local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensation reduction | Measurements will be recorded before drug injection and immediately after laceration repair.
  Participants will rate their sensation level on a visual analog scale from 0 to 10 both before the drug injection and after the laceration repair procedure. 0 indicating no sensation and 10 indicating worst sensation. Reduction in sensation will be calculated as the difference between the pre-injection and post-procedure sensation, with a larger number indicating a greater reduction in sensation.

SECONDARY OUTCOMES:
Anesthesia satisfaction by patient | Immediately after laceration repair
  Patient satisfaction of anesthesia yes/no
Anesthesia satisfaction by physician | Immediately after laceration repair
  Physician satisfaction of anesthesia yes/no

CONTACTS AND LOCATIONS:
Locations (1):
- Bethesda Hospital East, Boynton Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No